CLINICAL TRIAL: NCT01596517
Title: Efficacy and Effectiveness of Combination Therapy With Pegylated Interferon Alfa-2a and Ribavirin in Korean Patients With Chronic Hepatitis C
Brief Title: Efficacy and Effectiveness of PegInterferon and Ribavirin in Korean Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Severance Hospital (Other); Gangnam Severance Hospital (Other); Seoul St. Mary's Hospital (Other); Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Young-Suk Lim, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2003-0059
Record Dates: First submitted 2012-05-07; First posted 2012-05-11 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Korean CHC (Experimental): Two CHC patient groups. One is CHC patients who are treated with combination of peginterferon alfa-2a and ribavirin in a prospective, multicenter, industry-sponsored, open-label, uncontrolled, community-based clinical trial (Pegasys Expanded Access Program) conducted at 6 tertiary referral centers in Korea between 2003 and 2004. Another is a cohort of hepatitis C patients who were treated in a single tertiary referral hospital (Asan Medical Center, Seoul, Korea) between 2004 and 2008.
  Interventions: Drug: Peginterferon alfa-2a plus ribavirin for HCV genotype 1; Drug: Peginterferon alfa-2a plus ribavirin for HCV genotype 2/3

INTERVENTIONS:
Drug: Peginterferon alfa-2a plus ribavirin for HCV genotype 1 — Patients with genotype 1: treatment with peginterferon α-2a (Roche, Basel, Switzerland) 180 μg/week and daily ribavirin dose of 1,000 mg (for patients with body weight <75kg) or 1,200 mg (for patients with body weight ≥75kg) for 48 weeks.
  Other Names: Pegasys; Copegus
Drug: Peginterferon alfa-2a plus ribavirin for HCV genotype 2/3 — Patients with genotype 2 or 3: treatment with peginterferon α-2a 180 μg/week and daily ribavirin dose of 800 mg for 24 weeks.
  Other Names: Pegasys; Copegus

SUMMARY:
The purpose of this study is to investigate the efficacy and effectiveness of peginterferon alfa-2a and ribavirin therapy in Korean chronic hepatitis C patients.

DETAILED DESCRIPTION:
A retrospective analysis of a prospective, multicenter, industry-sponsored, open-label, uncontrolled, community-based clinical trial of combination of peginterferon alfa-2a and ribavirin (Pegasys Expanded Access Program) conducted at 6 tertiary referral centers in Korea between 2003 and 2004 and a cohort of hepatitis C patients who were treated in a single tertiary referral hospital (Asan Medical Center, Seoul, Korea) between 2004 and 2008

ELIGIBILITY:
Inclusion Criteria: all of below

* adults aged 18-70 years
* serum anti-HCV antibody (+)
* HCV RNA detectable by PCR
* compensated liver disease (Child-Pugh class A)

Exclusion Criteria: any of below

* HCV genotype other than 1, 2, or 3
* acute hepatitis C
* decompensated cirrhosis or hepatocellular carcinoma
* other liver disease such as hepatitis A or B, or autoimmune hepatitis
* HIV Ab(+)
* severe depression or other psychiatric disease
* previous organ transplantation
* absolute neutrophil count (ANC) < 1,000 cells/mm3 or platelet count < 75,000 cells/mm3, or hemoglobin (Hb) < 13 g/dL for men, <12 g/dL for women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2003-06; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving sustained virological response (SVR) | at 24 weeks after cessation of treatment
  SVR is defined as a documented undetectable serum HCV RNA by PCR at 24 weeks after cessation of treatment

SECONDARY OUTCOMES:
The proportion of patients achieving early virological response (EVR) | at 12 weeks of treatment
  EVR is defined as reduction of HCV RNA level by 2 log or more at 12 weeks of treatment
the proportion of patients achieving complete EVR (cEVR) | at 12 weeks of treatment
  cEVR is defined as HCV RNA undetectable by PCR at 12 weeks of treatment
The proportion of patients achieving end-of-treatment response (ETR) | at week 48 for HCV genotype 1 and at week 24 for HCV genotype 2/3
  ETR is defined as HCV RNA undetectable at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Heo NY, Lim YS, Lee HC, Lee YS, Kim KM, Byun KS, Han KH, Lee KS, Paik SW, Yoon SK, Suh DJ. High effectiveness of peginterferon alfa-2a plus ribavirin therapy in Korean patients with chronic hepatitis C in clinical practice. Clin Mol Hepatol. 2013 Mar;19(1):60-9. doi: 10.3350/cmh.2013.19.1.60. Epub 2013 Mar 25. PMID 23593611